CLINICAL TRIAL: NCT01734083
Title: The Effects of Whole Body Vibration Exercise Training on Physical Functioning and Falls in Community-dwelling Elderly With Cognitive Impairments
Brief Title: Whole Body Vibration Exercise for Elderly With Cognitive Impairments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Marco Yiu-Chung Pang, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20120929006
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Dementia
Keywords: rehabilitation; exercise; fall; muscle; vibration; mobility; cognition
MeSH Terms: conditions — Dementia; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Whole body vibration exercise (Experimental): The experimental group will receive 2 sessions of whole body vibration exercise training and conventional exercise per week for a period of 9 weeks. The total duration of vibration exposure per session will range from 4 to 6 minutes. The vibration frequency and amplitude used will be 30 Hz and 1 mm, respectively.
  Interventions: Device: Whole body vibration exercise; Behavioral: Conventional exercise
- Conventional exercise (Active Comparator): This group will receive 2 sessions of conventional exercise training per week for a period of 9 weeks.
  Interventions: Behavioral: Conventional exercise

INTERVENTIONS:
Device: Whole body vibration exercise — The whole body vibration will be delivered by a platform that can generate vibration signals (Powerplate). The total duration of vibration exposure per session will range from 4 to 6 minutes. The vibration bouts (30-45 seconds per bout) will be interspersed with a 1 to 2 minutes of rest period. While standing on the vibration platform, subjects will be instructed to repeat two exercises: (1) static semi-squats, and (2) dynamic semi-squats.
  Arms: Whole body vibration exercise
Behavioral: Conventional exercise — The conventional exercise training will involve a combination of upper limb and lower limb stretching and strengthening exercises, balance training, and gait re-education.

SUMMARY:
The whole body vibration exercise group will have significantly more improvement in mobility, muscle strength, balance, balance confidence, and cognitive function with a lower fall rate than the control group.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of mild or moderate dementia, with a Clinical Dementia Rating (CDR) of 1 to 2, and a Cantonese Mini-mental State Examination (CMMSE) score at 10 or above but below the local cutoff for dementia (18-22, depending on education level)
* able to stand for at least 1 minute with or without hand support
* living in the community
* having an informed consent (from the primary caregiver)

Exclusion Criteria:

* significant musculoskeletal conditions (e.g. amputations)
* metal implants in the lower extremity
* recent fracture in the lower extremity
* vestibular disorders
* peripheral vascular disease
* other serious illnesses or contraindications to exercise.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2012-11; Primary Completion 2015-01 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Timed-up-and-go test | week 0
  A measure of functional mobility
Timed-up-and-go test | week 9
Timed-up-and-go test | week 21

SECONDARY OUTCOMES:
Berg balance scale | week 0
Berg balance scale | week 9
Berg balance scale | week 21
Activities-specific balance confidence scale | week 0
Activities-specific balance confidence scale | week 9
Activities-specific balance confidence scale | week 21
five times sit-to-stand test | week 0
five times sit-to-stand test | week 9
five times sit-to-stand test | week 21
Mini-Mental State Examination | week 0
Mini-Mental State Examination | week 9
Mini-Mental State Examination | week 21
Quality of Life in Alzheimer's disease | week 0
Quality of Life in Alzheimer's disease | week 9
Quality of Life in Alzheimer's disease | week 21
incidence of falls | daily starting from week 0 to week 33
  Incidence of falls will be recorded by using fall diaries.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Pang, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Jockey Club Centre for Positive Ageing, Shatin, New Territories, Hong Kong

REFERENCES:
- [Background] Bautmans I, Van Hees E, Lemper JC, Mets T. The feasibility of Whole Body Vibration in institutionalised elderly persons and its influence on muscle performance, balance and mobility: a randomised controlled trial [ISRCTN62535013]. BMC Geriatr. 2005 Dec 22;5:17. doi: 10.1186/1471-2318-5-17. PMID 16372905
- [Background] Bruyere O, Wuidart MA, Di Palma E, Gourlay M, Ethgen O, Richy F, Reginster JY. Controlled whole body vibration to decrease fall risk and improve health-related quality of life of nursing home residents. Arch Phys Med Rehabil. 2005 Feb;86(2):303-7. doi: 10.1016/j.apmr.2004.05.019. PMID 15706558